CLINICAL TRIAL: NCT03358355
Title: Unacylated Ghrelin to Improve FuncTioning in PAD: The GIFT Trial
Acronym: GIFT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00202400
Record Dates: First submitted 2017-06-19; First posted 2017-11-30 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Artery Disease; PAD; Peripheral Arterial Disease
Keywords: PAD; unacylated ghrelin; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Subcutaneous injection of unacylated ghrelin: Doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg
  Interventions: Drug: unacelyated ghrelin

INTERVENTIONS:
Drug: unacelyated ghrelin — We will test doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg of unacylated ghrelin on three separate days for each participant.

SUMMARY:
The GIFT pilot study will investigate the optimal subcutaneous dose and safety of subcutaneously administered unacylated ghrelin in older people with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The pilot GIFT Trial will obtain preliminary evidence to identify the optimal dose of subcutaneously administered unacylated ghrelin in people with PAD. The results of this pilot study may be used to design a randomized trial of unacylated ghrelin, in subsequent study, to improve functioning and prevent mobility loss in older people with PAD.

In our primary specific aims, we will 1) establish the association of increasing doses of subcutaneous unacylated ghrelin with circulating levels of unacylated ghrelin 2) assess the safety of increasing doses of subcutaneously administered unacylated ghrelin in six patients with PAD age 55 and older. We will relate peak and Area Under the Curve values of unacylated ghrelin to brachial artery flow-mediated dilation (FMD) values. To achieve these aims, six PAD participants age 55 and older will receive a single subcutaneous injection of unacylated ghrelin at doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg, respectively, on three separate days at least one week apart. Unacylated ghrelin levels will be measured at baseline and at defined intervals after each subcutaneous injection (30 minutes, 60 minutes, 1.5 hours, 3 hours, 6 hours, 8 to 12 hours and 24 hours). Brachial artery FMD will be measured at baseline, before the unacylated ghrelin injection, approximately six hours, and 24 hours after each unacylated ghrelin injection. Blood will be collected and stored for potential later analyses of circulating biomarkers, such as inflammatory biomarkers.

This is a Phase I study to guide dose finding for a pilot study of unacylated ghrelin in people with PAD.

ELIGIBILITY:
Inclusion Criteria:

1. PAD patients age 55 and older

Exclusion Criteria:

1. Above or below-knee amputation, critical limb ischemia, and wheelchair confinement.
2. Cardiovascular event during the previous three months. [Note: Participants who have undergone coronary revascularization for a cardiac event during the previous three months may still qualify.]
3. Major medical illnesses including renal disease requiring dialysis, or cancer requiring treatment in the previous year.
4. Participation in another clinical trial or completion of a clinical trial in the previous month, unless they were in the control group of the previous trial.
5. Unwilling to attend nine study visits over approximately six months.
6. Surgery including lower extremity revascularization or orthopedic surgery in the previous month or anticipated surgery in the next three months.
7. Greater than 15 mmHg difference in blood pressure in both arm pressure measurements during the ankle brachial index (ABI), diagnosis of Raynaud's phenomenon, or unable to have the blood pressure checked in both arms.
8. Blood pressure < 90/50 at baseline.
9. Non-English speaking, a visual impairment that limits ability to read the consent, or a hearing impairment that interferes with study participation.
10. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Unacylated Ghrelin Intervention: Subcutaneous injection of unacylated ghrelin: Doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg
  unacelyated ghrelin: We will test doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg of unacylated ghrelin on three separate days for each participant.
Period: Overall Study
Arm/Group | Unacylated Ghrelin Intervention
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Ankle-Brachial Index (ABI) [Mean (Standard Deviation); unit: ratio] — The ABI measures systolic blood pressures in the right brachial, dorsalis pedis, and posterior tibial arteries and left dorsalis pedis, posterior tibial, and brachial arteries. Each measurement is performed twice. The ABI is calculated by dividing mean systolic pressures in each leg by the mean of the 4 brachial pressures.
  ratio | 0.69 (0.13)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (4.6)
Six-minute walk distance [Mean (Standard Deviation); unit: feet] | 1254.6 (531.8)

OUTCOME MEASURES:

1. Primary Outcome: Levels of Unacylated Ghrelin
Description: Levels of unacylated ghrelin are measured before and after every injection
Time Frame: Baseline and at scheduled intervals up to 24 hours after baseline
Population: Data originate from participants that received the injection and of which had data available
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Intervention(10 ug/kg): Subcutaneous injection of unacylated ghrelin: Doses of 10 ug/kg
  unacelyated ghrelin: We will test doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg of unacylated ghrelin on three separate days for each participant.
- Intervention(20 ug/kg): Subcutaneous injection of unacylated ghrelin: Doses of 20 ug/kg
  unacelyated ghrelin: We will test doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg of unacylated ghrelin on three separate days for each participant.
- Intervention(40 ug/kg): Subcutaneous injection of unacylated ghrelin: Doses of 40 ug/kg
  unacelyated ghrelin: We will test doses of 10 ug/kg, 20 ug/kg, and 40 ug/kg of unacylated ghrelin on three separate days for each participant.
Arm/Group | Intervention(10 ug/kg) | Intervention(20 ug/kg) | Intervention(40 ug/kg)
Number analyzed (Participants) | 5 | 6 | 4
pg/ml
  unacylated ghrelin level - Pre | 71.34 (58.67) | 58.01 (29.98) | 59.96 (31.34)
  unacylated ghrelin level - 30 min | 845.57 (300.12) | 1522.36 (1339.83) | 1102.99 (595.46)
  unacylated ghrelin level - 60 min | 772.33 (342.00) | 1719.38 (2012.57) | 1033.50 (623.85)
  unacylated ghrelin level - 90 min | 763.39 (446.80) | 1998.58 (3043.75) | 982.61 (584.37)
  unacylated ghrelin level - 180 min | 596.44 (371.88) | 900.83 (1078.23) | 694.51 (389.81)
  unacylated ghrelin level - 360 min | 373.09 (311.77) | 492.23 (489.99) | 410.49 (323.12)
  unacylated ghrelin level - 720 min | 240.94 (135.65) | 304.62 (294.16) | 339.46 (295.43)
  unacylated ghrelin level - 1440 min | 67.29 (48.64) | 57.30 (27.34) | 62.28 (34.03)

2. Secondary Outcome: Brachial Artery Flow-mediated Dilation (FMD)
Description: Brachial artery flow-mediated dilation in response to hyperemia. The outcome is reporting the MAX Relative FMD 60/90 (%), which is calculated as the highest FMD between the RH60 and RH90 results, as a percent.
Time Frame: Baseline, 6-8 hours after baseline, 24 hours after baseline.
Population: Data originate from participants that received the injection and of which had data available
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Intervention(10 ug/kg) | Intervention(20 ug/kg) | Intervention(40 ug/kg)
Number analyzed (Participants) | 5 | 5 | 6
ratio
  Change in FMD 60/90 (%) from baseline to 6 hours | 0.23 [-0.47 to 2.21] | 0.85 [0.63 to 1.17] | 0.06 [-1.56 to 1.67]
  Change in FMD 60/90 (%) from baseline to 24-hours | 1.14 [0.99 to 1.94] | -2.23 [-2.70 to -2.07] | 0.11 [-0.83 to 0.55]

3. Other Pre Specified Outcome: Number of Participants Who Experienced Adverse Events
Description: Adverse events
Time Frame: Within 24 hours after subcutaneous injection.
Population: Data originate from participants that received the injection and of which had data available
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention(10 ug/kg) | Intervention(20 ug/kg) | Intervention(40 ug/kg)
Number analyzed (Participants) | 5 | 6 | 6
Participants
  New swelling | 0 | 0 | 0
  New lightheadedness or dizziness | 0 | 1 | 0
  New headaches | 0 | 1 | 0
  New symptoms | 0 | 1 | 0

4. Other Pre Specified Outcome: Number of Participants Who Experienced Serious Adverse Events
Description: Serious adverse events
Time Frame: Within 24 hours after subcutaneous injection.
Population: Data originate from participants that received the injection and of which had data available
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored continuously throughout the study and will be reported to the DSMB and IRB in a timely manner according to pre-specified requirements. We will minimize risk by observing study participants for approximately 8-12 hours after each of the three doses of unacylated ghrelin.
Description: Participant that received any injection were monitored for adverse events.
Arm/Group | Intervention(10 ug/kg) | Intervention(20 ug/kg) | Intervention(40 ug/kg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention(10 ug/kg) (N=6) | Intervention(20 ug/kg) (N=6) | Intervention(40 ug/kg) (N=6)
Cardiovascular event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention(10 ug/kg) (N=6) | Intervention(20 ug/kg) (N=6) | Intervention(40 ug/kg) (N=6)
New swelling (General disorders) | 0 (0) | 0 (0) | 0 (0)
New lightheadedness or dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
New headaches (General disorders) | 0 (0) | 1 (1) | 0 (0)
New symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT03358355/Prot_SAP_000.pdf